CLINICAL TRIAL: NCT02052180
Title: Bupivicaine Extended-Release Liposome Injection Versus Marcaine for Early Post-Operative Pain Control Following Wrist Operations
Brief Title: Early Post-Operative Pain Control Following Wrist Operations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BVM-3-27
Record Dates: First submitted 2014-01-22; First posted 2014-01-31 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Pain
Keywords: Carpalmetacarpal arthroplasty; Proximal row carpectomy; Post-operative pain control; Exparel; Marcaine
MeSH Terms: conditions — Pain | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exparel (Experimental): EXPAREL arm: one vial (266 mg/20 mL) of EXPAREL (Bupivicaine Extended-Release Liposome, 13.3mg/ml), undiluted, will be administered for each of the specified procedures.
  Interventions: Drug: Exparel
- Control (Active Comparator): 15 cc of Marcaine 0.5% (Bupivacaine 0.5%, 5mg/ml) will be administered into the wrist per the Surgeon's Standard practice.
  Interventions: Drug: Marcaine (Control)

INTERVENTIONS:
Drug: Exparel — EXPAREL arm: one vial (266 mg/20 mL) of EXPAREL (Bupivicaine Extended-Release Liposome, 13.3mg/ml), undiluted, will be administered for each of the specified procedures.
  Arms: Exparel
Drug: Marcaine (Control) — 15 cc of Marcaine 0.5% (Bupivacaine 0.5%, 5mg/ml) will be administered into the wrist per the Surgeon's Standard practice.
  Arms: Control

SUMMARY:
The purpose of this study is to demonstrate improved pain control and outcomes in wrist operations with the use of a long-acting local anesthetic, EXPAREL, when compared to the use of the standard local anesthetic, Marcaine.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* ASA physical status 1-3
* Undergoing either carpometacarpal arthroplasty or proximal row carpectomy operation
* Physically and mentally able to participate in the study and complete all study assessments
* Able to voluntarily give fully informed consent to participate in this study and complete all study assessments within the timeframes required.

Exclusion Criteria:

* History of hypersensitivity or idiosyncratic reactions to amide-type local anesthetics
* Any patient whose anatomy, or surgical procedure, in the opinion of the Investigator, might preclude the potential successful local administration of EXPAREL
* Patients who have received any investigational drug within 30 days prior to EXPAREL administration, or planned administration of another investigational product or procedure during their participation in this study
* Any chronic condition requiring use of opioids for treatment of the medical condition for three (3) months or more
* Confirmed pregnancy at time of enrollment
* Patients unable to comply with the study requirements, i.e. inaccessible by phone, or deaf

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Changes in Pain | Pre-op, Post-op days: 1,2,3,4, and 14
  Pain measured by Numeric Rating Scale (NRS)

CONTACTS AND LOCATIONS:
Overall Officials: Jason P. Rehm, MD, Principal Investigator — University of Tennessee College of Medicine Chattanooga
Locations (1):
- UTCOM Chattanooga Department of Plastic Surgery, Chattanooga, Tennessee, United States